CLINICAL TRIAL: NCT01044667
Title: Reduced Gastrointestinal Complaints and Improved Quality of Life in Lung Transplant Recipients Converted From Mycophenolate Mofetil (MMF) to Myfortic (Enteric-coated Mycophenolate Sodium, Ec-mps)
Brief Title: A Gastrointestinal Quality of Life Study in Lung Transplant Recipients Converted From Mycophenolate Mofetil to Myfortic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment and lack of study staff
Sponsor: Vanderbilt University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Myfortic 091423
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients taking Myfortic (Other): Lung transplant patients converted from MMF to Myfortic as part of standard of care treatment will have GI and Quality of Life assessments done at the time of conversion to Myfortic and at 60 days, 90 days and 180 days.
  Interventions: Behavioral: GI and Quality of Life Assessment

INTERVENTIONS:
Behavioral: GI and Quality of Life Assessment

SUMMARY:
The primary objective of this study is to evaluate gastrointestinal (GI) symptoms and health related quality of life in lung transplant recipients converted from Mycophenolate Mofetil (MMF) to Myfortic as part of standard immunosuppressive therapy.

DETAILED DESCRIPTION:
Subjects administered MMF as part of their immunosuppression regimen after lung transplantation have a high incidence of GI symptoms related to the known side-effects of this drug. Previous studies have shown that GI symptoms are an important predictor of health related quality of life in other solid organ transplants (1). GI complications are common after lung transplant (2). We hypothesize that lung transplant patients converted from MMF to Myfortic will have significant reduction in severity of GI complaints. We also hypothesize that improvement in the severity of GI complaints will lead to an improved quality of life in these subjects. The study also includes data to evaluate the effect of GI complaints on health related quality of life.

Patients will complete questionnaires at each visit. Calls from the patients to the lung transplant center with GI complaints will be queried and documented on the case report form by the research nurse at each study visit. Similarly, hospital admissions for GI related complaints in the cohort will be documented. Symptom severity and health related quality of life will be assessed through the following questionnaires that have previously been validated in populations other than lung transplant (1). These questionnaires are selected specifically to capture the impact of GI complaints as related to the health related quality of life. The questionnaires that will be completed by the patient:

i.Gastrointestinal Quality of Life Index (GIQLI)

• The GIQLI is a 36-item questionnaire that assess the impact of GI distress on daily life

ii.SF-36 Health Survey • "The SF-36 Health Survey is a questionnaire that capture practical, reliable, and valid information about functional health and well-being from the patients' point of view" (4)

iii.EQ-5D Health Questionnaire

• "The EQ-5D is a standardized instrument for use as a measure of health outcome. The EQ-5D provides a simple descriptive profile and a single value for health status" (5)

Patients will complete the three questionnaires at 4 outpatient visits occurring:

* when the patient comes in to an outpatient clinic visit after initial hospital discharge after lung transplantation with complaints of GI distress (Day 1-Convert to Myfortic);
* 60 Days;
* 90 days;
* 180 days

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent and adhere to study regimen
* Recipients who are 18-70 years of age
* Patients who have undergone either single or double lung transplant are discharged on the standard MMF (no generic MMF will be used) therapy and complain of GI symptoms, thought to be related to their immunosuppressive regimen

Exclusion Criteria:

* Patients who have GI complaints thought to be due to factors other than immunosuppressive regimen
* Patients receiving steroid treatment for acute rejection
* Women of childbearing potential who do not agree to use at least two acceptable forms of contraception prior to starting study drug, while taking study drug, and for 6 weeks after stopping study drug
* Women who have a positive serum or urine pregnancy test at visit 1 and/or continuing through the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal Quality of Life Index (GIQLI), Baseline to 60 days: | Change from Baseline to 60 days
  Change in GIQLI after conversion from MMF to Myfortic
Change in SF-36 Health Survey, Baseline to 60 days | Change from Baseline to 60 days
  Change in SF-36 Health Survey after conversion from MMF to Myfortic
Change in EQ-5D Health Questionnaire, Baseline to 90 days | Change from Baseline to 60 days
  Change in EQ-5D Health Questionnaire after conversion from MMF to Myfortic

SECONDARY OUTCOMES:
Gastrointestinal Quality of Life Index (GIQLI) | Day 90 and Day 180
  Change in GIQLI after conversion from MMF to Myfortic
SF-36 Health Survey | Day 90 and Day 180
  Change in SF-36 Health Survey after conversion from MMF to Myfortic
EQ-5D Health Questionnaire | Day 90 and Day 180
  Change in EQ-5D Health Questionnaire after conversion from MMF to Myfortic

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lambright, MD, Principal Investigator — Vanderbilt University Medcial Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States